CLINICAL TRIAL: NCT01228370
Title: A 12-week, Open-label, Multi-center Study to Evaluate the Clinical Efficacy and Safety of Silodosin on Voiding Dysfunction Associated With Neurogenic Bladder
Brief Title: Efficacy and Safety of Silodosin on Voiding Dysfunction Associated With Neurogenic Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWP-SDS-402
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Neurogenic Bladder; Voiding Dysfunction
Keywords: sildosin; neurogenic bladder; voiding dysfunction
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silodosin (Experimental): Silodosin 8mg once a day for 12 weeks
  Interventions: Drug: silodosin

INTERVENTIONS:
Drug: silodosin — silodosin 8mg once a day for 12 weeks

SUMMARY:
Because the bladder neck and proximal urethra contain abundant α1-adrenergic receptors, α-blockers or α1-blockers are well-known to reduce bladder neck obstruction in patients with or without neurogenic bladder.

α1-blockers seem to have a potential to reduce bladder outlet resistance during voiding in patients with neurogenic bladder.

Based on these turnouts, we designed this clinical study to evaluate the clinical effect and safety of silodosin on voiding dysfunction associated with neurogenic bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is 20 years old or over
* Patient who is diagnosed with neurogenic bladder through urodynamic test, having urinary disorder symptoms
* In case, patient has been taking concomitant drugs allowed for the study, only if the doses have been stable within 8 weeks from the screening visit
* Patient who has a I-PSS score of 8 or over
* Patient who has a QoL score of 3 or over
* Patient who has a Qmax of below 15 mL/sec
* Patient who has a PSA<4.0 ng/mL or has PSA>4.0 ng/mL with no opinion of prostate cancer from biopsy
* Patient who is willing to take the investigational product in accordance with the protocol
* Patient who is able to fill out questionnaire and understand requirements of the study including informed consent
* Patient voluntarily decides to participate and signs the written consent form.

Exclusion Criteria:

* Patient who hs urinate at all on his/her own.
* Patient who has a history of bladder surgery
* Patient who has detrusor areflexia or acontractile bladder diagnosed by urodynamic test
* Patient who has a postvoid residual urine volume(PRV) of 300 mL or greater, or has a PRV of 50% or over of the maximum bladder capacity
* Patient who has a prostate volume of 30 mL or greater resulted from a severe benign prostatic hyperplasia(BPH) (only in case of male)
* Patient who has urethral stricture
* Patient who has symptomatic urinary tract infection(UTI) before screening visit
* Patient who has a gross hematuria(except idiopathic hematuria)
* Patient who conducts Clean Intermittent Catheterization(CIC)
* Patient who has been taking α-blocker other than silodosin or α-agonist within 8 weeks from screening visit
* Patient who has a Botulinum toxin injection for bladder problems within at least 1 year from screening visit
* Patient who has severe hapatic disorders(hepatic insufficiency, cirrhosis, jaundice, hepatoma)or has a total bilirubin of 2.5 mg/dL or higher or has AST/ALT 2.5 times higher than the normal upper limit
* Patient who has a renal impairment with a serum creatinine 2.0 mg/dL or higher
* Patient who has experienced severe arrhythmia, cardiac failure, myocardiac infarction, unstable angina, cerebral infarction within 6 months from screening visit
* Patient who has orthostatic hypotention before screening visit
* Patient who has a demanding chronic disease
* Patient who has an allergy to drugs
* Patient who is prohibited from taking silodosin
* Patient who has to take drugs prohibited from the study during the clinical study
* Patient who is pregnant or plans to be pregnant or is breastfeeding or is not practicing contraception using medically acceptable contracenption
* Patient who has experienced any other clinical study within 4 weeks from screening visit
* Patient who is excluded from medical dicisions made by the investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
I-PSS score change after treatment | 12 weeks

SECONDARY OUTCOMES:
Change in Qmax after treatment | 12 weeks
Change in Postvoid Residual urine Volume(PRV) after treatment | 12 weeks
Change in I-PSS Quality of Life after treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Yoon Kim, Principal Investigator — Daegu Catholic University Medical Center; Chul-Hee Park, Principal Investigator — Keimyung Univ. Dongsan Medical Center; Hee-Chang Jung, Principal Investigator — Yeungnam Univ. Medical Center; Kyung-Hyun Moon, Principal Investigator — Ulsan Univ. Hospital; Tae-Hee Oh, Principal Investigator — Samsung Changwon Hospital; Jae-Soo Kim, Principal Investigator — Daegu Fatima Hospital
Locations (6):
- South Korea (6):
  - Daegu Catholic Univ. Medical Center, Daegu, Daegu City
  - Daegu Fatima Hospital, Daegu, Daegu City
  - Keimyung Univ. Dongsan Medical Center, Daegu, Daegu City
  - Yeungnam Univ. Medical Center, Daegu, Daegu City
  - Samsung Changwon Hospital, Changwon, Gyeongsangnam-do
  - Ulsan Univ. Hospital, Ulsan, Ulsan City